CLINICAL TRIAL: NCT03708315
Title: Safety and Efficacy of BXCL501, a Sublingual Film Delivery of Dexmedetomidine for the Treatment of Acute Agitation in Schizophrenia
Brief Title: BXCL501 for Agitation in Schizophrenia
Acronym: DEX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000023998
Record Dates: First submitted 2018-10-12; First posted 2018-10-17 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: The subjects will be randomized and will get either a sublingual formulation of dexmedetomidine or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Order 1 (Active Comparator): Subjects will be given a sublingual formulation of BXCL501 (dexmedetomidine)
  Interventions: Drug: Dexmedetomidine Hydrochloride
- Order 2 (Placebo Comparator): Subjects will be given a sublingual film of placebo.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — Dexmedetomidine Hydrochloride
  Other Names: Precedex
  Arms: Order 1
Drug: Placebos — Placebo
  Arms: Order 2

SUMMARY:
Agitation is characterized by excessive motor or verbal activity, irritability, uncooperativeness, threatening gestures, and, in some cases, aggressive or violent behavior. While agitation may have various underlying causes, patients with schizophrenia are especially vulnerable to acute episodes of agitation, especially during exacerbation of disease, and clinicians do not always diagnose these episodes early enough. Agitation associated with psychosis is a frequent reason for emergency department visits, and unless it is recognized early and managed effectively, it can rapidly escalate to potentially dangerous behaviors, including physical violence. Educating psychiatric professionals about the timely and accurate diagnosis of agitation among patients with schizophrenia or bipolar disorder and developing a well-tolerated easily administered medication will contribute to the prompt and effective management of this condition and could help reduce the risk of violent behavior and other undesirable outcomes. This study is designed to identify the ideal dose range and tolerability of sublingual Dexmedetomidine in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give informed consent.
2. Male or female between 18 and 65 years of age, inclusive
3. According to DSM-V meet criteria for Schizophrenia or Schizoaffective disorder.

Exclusion Criteria:

1. Current significant medical condition or other comorbidities
2. Current substance dependence
3. Women who are pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Symptom Scale Excited Component (PANSS-EC) | Measured at screening, prior to dosing, every 30 minutes post drug administration, and the day following drugadministration.
  PANSS-EC comprises 5 items associated with agitation: poor impulse control, tension, hostility, uncooperativeness, and excitement; each scored from 1 (minimum) to 7 (maximum). The PANSS-EC is the sum of these 5 subscales and ranges from 5 to 35.
Skin conductance response (SCR) | Measured continuously from approximatley 15 minutes prior to drug administatration until the end of the test day (approximately 11 hours)
  SCR is one of the fastest-responding measures of stress response and arousal. Along with changes in heart rate, it has been found to be one of the most robust and non-invasive physiological measures of autonomic nervous system activity.
Heart rate variability | Measured continuously from approximatley 15 minutes prior to drug administatration until the end of the test day (approximately 11 hours)
  Heart rate variability (HRV) is a measure of the variability in time intervals between heart beats and is sensitive to sympathetic activity as well as worsening of psychosis/agitation.
Blood pressure | Measured at screening, prior to administartion, approximately every 15 minutes post drug administration, and one day after drug administration
  Systolic and diastolic blood pressure
Agitation-Calmness Scale (ACES) | Measured at screening, prior to administration, approximately every 30 minutes post dose, and one day following drug administration.
  Designed to assess the clinical levels of calmness and sedation. This is a 9-point scale that differentiates between agitation, calmness, and sleep states Scores range from 1 (marked agitation)-9 (unarousable).
Richmond Agitation Sedation Scale (RASS) | Measured at screening, prior to administration, approximately every 30 minutes post dose, and one day following drug administration.
  The RASS is a 10-level rating scale ranging from "Combative" (+4) to "unarousable" (-5).

SECONDARY OUTCOMES:
Behavioral Activity Rating Scale (BARS) | Measured at screening, prior to administration, approximately every 30 minutes post dose, and one day following drug administration.
  Ranging from 1 to 7 where: 1 = difficult or unable to rouse, 2 = asleep but responds normally to verbal or physical contact, 3 = drowsy, appears sedated, 4 = quiet, and awake (normal level of activity), 5 = signs of overt (physical or verbal) activity, calms down with instructions, 6 = extremely or continuously active, not requiring restraint, 7 = violent, requires restraint.
Clinical Global Impressions-Improvement Scale (CGI-I) | Measured at screening, prior to dosing, every 30 minutes post drug administration, and the day following drugadministration.
  Clinical Global Impression- Improvement (CGI-I) scores ranged from 1 to 7: 0=not assessed (missing), 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse.
Adverse Effects | Assessed prior to dosing, throughout study drug administration, and up to one week after drug administration
  To determine any adverse effects on blood pressure, heart rate, or respiratory drive occurs before or coincident with the achievement of the aforementioned level of sedation.

CONTACTS AND LOCATIONS:
Overall Officials: Mohini Ranganathan, MD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States